CLINICAL TRIAL: NCT00657384
Title: Tranexamic Acid Versus Placebo to Reduce Perioperative Bleeding After Major Hepatectomy : a Prospective Randomized Double-blinding Study
Brief Title: Tranexamic Acid Versus Placebo to Reduce Perioperative Bleeding After Major Hepatectomy
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 3959
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Blood Loss, Surgical
Keywords: Specify the primary condition or disease being studied Major Hepatectomy
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- acid tranexamic (Experimental): acid tranexamic
  Interventions: Drug: acid tranexamic
- 2 (Placebo Comparator): Nacl 0.9%
  Interventions: Drug: Nacl 0.9%

INTERVENTIONS:
Drug: acid tranexamic — 10 mg/kg Iv after randomization of the patient in the study,follow-up by continuous infusion of 10 mg/kg/h up to the end of the intervention.
  Arms: acid tranexamic
Drug: Nacl 0.9% — 10 mg/kg Iv after randomization of the patient in the study,follow-up by continuous infusion of 10 mg/kg/h up to the end of the intervention
  Arms: 2

SUMMARY:
Blood loss was reported as a prognostic risk factor of morbidity and overall survival after hepatic resection. The aim of this study prospective randomized was compare the efficacy of the administration of tranexamic acid versus placebo to reduce perioperative bleeding after major hepatectomy (> 3 hepatic segments).

ELIGIBILITY:
Inclusion Criteria:

* Signature of the consent form
* Patients with hepatic lesion needing a major hepatectomy (≥ 3 hepatic segments)

Exclusion Criteria:

* Absence of signature of the consent form
* Patient with cirrhosis
* Minor hepatectomy (< 3 hepatic segments)
* Hepatectomy associated with vascular resection
* Contraindication of tranexamic acid : history of arterial or venous thrombosis , disseminated intravascular coagulation, severe renal insufficiency, history of epilepsies , intrathecal or intraventricular injection
* Pregnant or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2008-08-20 (Actual); Primary Completion 2013-08-20 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The volume of compensated blood loss with the formula: [TBV x (initial hematocrit - final hematocrit ) + number of transfused RBC unit] with TBV=Total Blood Volume and RBC= red blood cell (1 RBC unit = 500 ml with hematocrit=30%). | at day 5

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Pessaux, Principal Investigator — CHU strasbourg
Locations (4):
- France (4):
  - CHU Amiens, Hôpital Nord, Amiens
  - Chirurgie digestive et transplantation, Hôpital de Besançon, Besançon
  - CHU de Bordeaux (Hôpital Haut- Lévêque et Hôpital Saint-André), Bordeaux
  - Chirurgie Viscérale et transplantation, Hôpital de Hautepierre , CHU Strasbourg, Strasbourg